CLINICAL TRIAL: NCT03021018
Title: A Multicenter, Open-Label, Randomized, Parallel-Group, Active-Controlled Study to Assess the Efficacy and Safety of Brivaracetam Administered Intravenously as Treatment for Increased Seizure Activity in an Epilepsy Monitoring Unit Setting
Brief Title: A Study to Assess the Efficacy and Safety of Brivaracetam as Treatment for Increased Seizure Activity in an Epilepsy Monitoring Unit Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EP0087
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Epilepsy
Keywords: Epilepsy; Brivaracetam; Epilepsy Monitoring Unit; Increased seizure activity
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam; Lorazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brivaracetam (BRV) 100 mg (Experimental): Two 5 ml vials of brivaracetam administered intravenously over a 2-minute period
  Interventions: Drug: Brivaracetam
- Brivaracetam (BRV) 200 mg (Experimental): Four 5 ml vials of brivaracetam administered intravenously over a 4-minute period
  Interventions: Drug: Brivaracetam
- Lorazepam (LZP) (Active Comparator): Lorazepam bolus is to be injected based on information from the patient leaflet/package insert. The rate of injection should not exceed 2.0 mg/min. The LZP dose will be determined according to the Investigator's clinical judgment.
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Brivaracetam — * Pharmaceutical Form: Solution for infusion
  * Concentration: 10 mg/ml
  * Route of Administration: intravenous
  Other Names: Briviact
  Arms: Brivaracetam (BRV) 100 mg; Brivaracetam (BRV) 200 mg
Drug: Lorazepam — * Pharmaceutical Form: Solution for injection
  * Route of Administration: intravenous
  Arms: Lorazepam (LZP)

SUMMARY:
The purpose of this study is to assess the efficacy of intravenous brivaracetam (BRV) compared to intravenous lorazepam (LZP) in subjects with epilepsy undergoing Epilepsy Monitoring Unit (EMU) evaluation who experience seizures that require prompt treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, 18 to 70 years of age, inclusive
* Subject has an established diagnosis of epilepsy
* Subject has been admitted to the institution's Epilepsy Monitoring Unit (EMU) for seizure characterization or noninvasive presurgical evaluation or such admission is planned within 21 days of Screening

Exclusion Criteria:

* Subject has previously participated in this study and was treated with study drug. Re-screen is permitted
* Subject has participated in another study of an investigational medicinal product (IMP) or a medical device within the previous 30 days of Epilepsy Monitoring Unit (EMU) admission or is currently participating in another study of an IMP or a medical device
* Subject has taken brivaracetam (BRV) in the 21 days prior to EMU admission
* History or presence of status epilepticus during the 6 months prior to EMU admission
* Subject has a medical or psychiatric condition that in the opinion of the Investigator could jeopardize or would compromise the subject's ability to participate in this study
* Subject has > 2x upper limit of normal (ULN) of any of the following: alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, or > ULN total bilirubin
* Subject has chronic liver disease
* Subject has hypersensitivity to BRV or any of its excipients
* Subject has a history of alcohol or drug abuse during the 6 months prior to EMU admission
* Subject with a history of psychogenic seizures
* Subject is a pregnant or lactating female
* Subject has a history of a significant Adverse Event (AE) due to a benzodiazepine in the opinion of the Investigator
* Subject has respiratory failure (or is at risk for respiratory failure), untreated sleep apnea, or other severe cardiorespiratory disease with New York Heart Association Class III or IV functional status, or requires supplemental oxygen
* Subject has acute narrow-angle glaucoma or myasthenia gravis
* Subject is receiving benzodiazepine treatment (defined as an average of >=4 administrations per week) that started less than 28 days prior to EMU admission
* Subject has a known allergic reaction or intolerance to benzodiazepines or benzodiazepine excipients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB (+1 844 599 2273)
Locations (14):
- United States (14):
  - Ep0087 108, Birmingham, Alabama
  - Ep0087 117, Tucson, Arizona
  - Ep0087 112, Orlando, Florida
  - Ep0087 115, Chicago, Illinois
  - Ep0087 113, Chicago, Illinois
  - Ep0087 119, Wichita, Kansas
  - Ep0087 116, Belmont, Massachusetts
  - Ep0087 106, Boston, Massachusetts
  - Ep0087 107, Detroit, Michigan
  - Ep0087 125, Lebanon, New Hampshire
  - Ep0087 120, Rochester, New York
  - Ep0087 121, Chapel Hill, North Carolina
  - Ep0087 105, Charlotte, North Carolina
  - Ep0087 123, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.clinicalstudydatarequest.com and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if a determination is made that the data cannot be adequately anonymized.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.clinicalstudydatarequest.com and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- See also: Product Information — http://www.briviact.com/briviact-PI.pdf?v=1479491757
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in February 2017 and concluded in April 2018.
Pre-assignment Details: Participant Flow refers to the Intent-to-Treat as Treated (ITT-T) Set.
Groups:
- Lorazepam (LZP): Lorazepam bolus was injected based on information from the patient leaflet/package insert. The lorazepam (LZP) dose was determined according to the Investigator's clinical judgment.
Period: Overall Study
Arm/Group | Lorazepam (LZP) | Brivaracetam (BRV) 100 mg | Brivaracetam (BRV) 200 mg
Started | 16 | 15 | 15
Completed | 14 | 15 | 15
Not Completed | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Fall with subsequent nasal fracture | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Intent-to-Treat as Treated Set which consisted of subjects who were treated with investigational medicinal product (IMP) regardless of qualifying seizure status.
Arm/Group | Lorazepam (LZP) | Brivaracetam (BRV) 100 mg | Brivaracetam (BRV) 200 mg | Total Title
Number analyzed (Participants) | 16 | 15 | 15 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 1
  Between 18 and 65 years | 16 | 14 | 13 | 43
  >=65 years | 0 | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.10 (11.18) | 43.92 (12.41) | 41.59 (15.98) | 42.18 (13.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 4 | 23
  Male | 5 | 7 | 11 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1 | 2
  Black or African American | 4 | 2 | 2 | 8
  White | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Time to Next Seizure (Per Clinical Observation With Electroencephalogram [EEG] Confirmation) or Rescue Medication
Description: This variable was calculated in hours. The event of next seizure was defined as the first seizure (clinically observed with electroencephalogram [EEG] confirmation) with the start date and time within 12 hours after the end of investigational medicinal product (IMP) administration.
Time Frame: During the Treatment Period (Day 1) until Safety Follow-Up Visit (Day 2)
Population: The Intent-to-Treat as Randomized (ITT-R) Set consisted of all randomized subjects who received the investigational medicinal product (IMP) for qualifying seizures.
Measure: Median (95% Confidence Interval); unit: hours
Groups:
- Lorazepam (LZP) (ITT-R): Lorazepam bolus was injected based on information from the patient leaflet/package insert. The LZP dose was determined according to the Investigator's clinical judgment. Subjects formed the Intent-to-Treat as Randomized (ITT-R) Set which consisted of all randomized subjects who received the investigational medicinal product (IMP) for qualifying seizures.
- Brivaracetam (BRV) 100 mg (ITT-R): Two 5 ml vials of brivaracetam administered intravenously over a 2-minute period. Subjects formed the ITT-R Set which consisted of all randomized subjects who received the investigational medicinal product (IMP) for qualifying seizures.
- Brivaracetam (BRV) 200 mg (ITT-R): Four 5 ml vials of brivaracetam administered intravenously over a 4-minute period. Subjects formed the ITT-R Set which consisted of all randomized subjects who received the investigational medicinal product (IMP) for qualifying seizures.
Arm/Group | Lorazepam (LZP) (ITT-R) | Brivaracetam (BRV) 100 mg (ITT-R) | Brivaracetam (BRV) 200 mg (ITT-R)
Number analyzed (Participants) | 15 | 15 | 15
hours | NA [5.55 to NA] — Due to the low numbers of events seen in the study, the Upper Confidence Limit (UCL) was not calculable. | NA [6.93 to NA] — Due to the low numbers of events seen in the study, the Upper Confidence Limit (UCL) was not calculable. | NA [4.33 to NA] — Due to the low numbers of events seen in the study, the Upper Confidence Limit (UCL) was not calculable.

2. Secondary Outcome: Time to Next Seizure (Per Clinical Observation) or Rescue Medication
Description: This variable was calculated in hours. The event of next seizure was defined as the first seizure (clinically observed and not necessarily confirmed via electroencephalogram [EEG]) with the start date and time within 12 hours after the end of investigational medicinal product (IMP) administration.
Time Frame: During the Treatment Period (Day 1) until Safety Follow-Up Visit (Day 2)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Lorazepam (LZP) (ITT-R) | Brivaracetam (BRV) 100 mg (ITT-R) | Brivaracetam (BRV) 200 mg (ITT-R)
Number analyzed (Participants) | 15 | 15 | 15
hours | NA [5.55 to NA] — Due to the low numbers of events seen in the study, the Upper Confidence Limit (UCL) was not calculable. | NA [6.93 to NA] — Due to the low numbers of events seen in the study, the Upper Confidence Limit (UCL) was not calculable. | NA [4.33 to NA] — Due to the low numbers of events seen in the study, the Upper Confidence Limit (UCL) was not calculable.

3. Secondary Outcome: Percentage of Subjects Who Are Seizure-free Per Clinical Observation at 6 Hours After the End of Study Drug Administration
Description: This variable was defined as the number of subjects seizure free during 6 hours after the end of study drug administration divided by the number of subjects in the Intent-to-Treat (ITT) set multiplied by 100.
Time Frame: At 6 hours after the end of study drug administration
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Lorazepam (LZP) (ITT-R) | Brivaracetam (BRV) 100 mg (ITT-R) | Brivaracetam (BRV) 200 mg (ITT-R)
Number analyzed (Participants) | 15 | 15 | 15
percentage of participants | 73.3 | 86.7 | 80.0

4. Secondary Outcome: Percentage of Subjects Who Are Seizure-free Per Clinical Observation at 8 Hours After the End of Study Drug Administration
Description: This variable was defined as the number of subjects seizure free during 8 hours after the end of study drug administration divided by the number of subjects in the ITT set multiplied by 100.
Time Frame: At 8 hours after the end of study drug administration
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Lorazepam (LZP) (ITT-R) | Brivaracetam (BRV) 100 mg (ITT-R) | Brivaracetam (BRV) 200 mg (ITT-R)
Number analyzed (Participants) | 15 | 15 | 15
percentage of participants | 73.3 | 80.0 | 80.0

5. Secondary Outcome: Percentage of Subjects Who Are Seizure-free Per Clinical Observation at 12 Hours After the End of Study Drug Administration
Description: This variable was defined as the number of subjects seizure free during 12 hours after the end of study drug administration divided by the number of subjects in the ITT set multiplied by 100.
Time Frame: At 12 hours after the end of study drug administration
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Lorazepam (LZP) (ITT-R) | Brivaracetam (BRV) 100 mg (ITT-R) | Brivaracetam (BRV) 200 mg (ITT-R)
Number analyzed (Participants) | 15 | 15 | 15
percentage of participants | 60.0 | 80.0 | 80.0

6. Secondary Outcome: Percentage of Subjects Who Receive Rescue Medication During the 6 Hours After the End of Study Drug Administration
Description: This variable was defined as the number of subjects who received rescue medication with start date and time within the first 6 hours after the end of study drug administration divided by the number of subjects in the Intent-to-Treat as randomized (ITT-R) set multiplied by 100.
Time Frame: During the 6 hours after the end of study drug administration
Population: as for outcome 1
Measure: Number; unit: percentage of participnats
Arm/Group | Lorazepam (LZP) (ITT-R) | Brivaracetam (BRV) 100 mg (ITT-R) | Brivaracetam (BRV) 200 mg (ITT-R)
Number analyzed (Participants) | 15 | 15 | 15
percentage of participnats | 20.0 | 0 | 6.7

7. Secondary Outcome: Percentage of Subjects Who Receive Rescue Medication During the 8 Hours After the End of Study Drug Administration
Description: This variable was defined as the number of subjects who received rescue medication with start date and time within the first 8 hours after the end of study drug administration divided by the number of subjects in the ITT-R set multiplied by 100.
Time Frame: During the 8 hours after the end of study drug administration
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Lorazepam (LZP) (ITT-R) | Brivaracetam (BRV) 100 mg (ITT-R) | Brivaracetam (BRV) 200 mg (ITT-R)
Number analyzed (Participants) | 15 | 15 | 15
percentage of participants | 26.7 | 6.7 | 13.3

8. Secondary Outcome: Percentage of Subjects Who Receive Rescue Medication During the 12 Hours After the End of Study Drug Administration
Description: This variable was defined as the number of subjects who received rescue medication with start date and time within the first 12 hours after the end of study drug administration divided by the number of subjects in the ITT-R set multiplied by 100.
Time Frame: During the 12 hours after the end of study drug administration
Population: as for outcome 1
Measure: Number; unit: percentage of participnats
Arm/Group | Lorazepam (LZP) (ITT-R) | Brivaracetam (BRV) 100 mg (ITT-R) | Brivaracetam (BRV) 200 mg (ITT-R)
Number analyzed (Participants) | 15 | 15 | 15
percentage of participnats | 40.0 | 6.7 | 13.3

ADVERSE EVENTS:
Time Frame: From Screening, at Day -28 and up to Safety Follow-Up (24 hours after the end of drug administration).
Groups:
- Lorazepam (LZP) (ITT-T): Lorazepam bolus was injected based on information from the patient leaflet/package insert. The LZP dose was determined according to the Investigator's clinical judgment. Subjects formed the Intent-to-Treat as Treated (ITT-T) Set which consisted of subjects who were treated with investigational medicinal product (IMP) regardless of qualifying seizure status.
- Brivaracetam (BRV) 100 mg (ITT-T): Two 5 ml vials of brivaracetam administered intravenously over a 2-minute period. Subjects formed the ITT-T Set which consisted of subjects who were treated with investigational medicinal product (IMP) regardless of qualifying seizure status.
- Brivaracetam (BRV) 200 mg (ITT-T): Four 5 ml vials of brivaracetam administered intravenously over a 4-minute period. Subjects formed the ITT-T Set which consisted of subjects who were treated with investigational medicinal product (IMP) regardless of qualifying seizure status.
Arm/Group | Lorazepam (LZP) (ITT-T) | Brivaracetam (BRV) 100 mg (ITT-T) | Brivaracetam (BRV) 200 mg (ITT-T)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 4/16 | 6/15 | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lorazepam (LZP) (ITT-T) (N=16) | Brivaracetam (BRV) 100 mg (ITT-T) (N=15) | Brivaracetam (BRV) 200 mg (ITT-T) (N=15)
Seizure cluster (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lorazepam (LZP) (ITT-T) (N=16) | Brivaracetam (BRV) 100 mg (ITT-T) (N=15) | Brivaracetam (BRV) 200 mg (ITT-T) (N=15)
Atrioventricular dissociation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT03021018/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT03021018/SAP_001.pdf